CLINICAL TRIAL: NCT02501850
Title: The Effect of the GLP-1 Receptor Agonists on Blood Levels of Lipoprotein (a)
Acronym: EGLIPA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VHI-GLP-2014-01
Record Dates: First submitted 2015-07-16; First posted 2015-07-17 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Lipoprotein (a)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Liraglutide; Exenatide; lixisenatide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Type 2 diabetic patients whom were prescribed GLP-1R agonists by the endocrinologist, according to usual clinical practice (liraglutide, exenatide, lixisenatide). The intervention is the prescription of an GLP-1R agonist (liraglutide, exenatide, lixisenatide)
  Interventions: Drug: Liraglutide
- Group B (Active Comparator): Type 2 diabetic patients whom were prescribed metformin and/or sulphonilurea, according to usual clinical practice.
  Interventions: Drug: metformin

INTERVENTIONS:
Drug: Liraglutide — Treatment with liraglutide, exenatide or lixisenatide
  Other Names: Exenatide; Lixisenatide
  Arms: Group A
Drug: metformin — Treatment with metformin and/or sulphonilurea
  Other Names: sulphonilurea
  Arms: Group B

SUMMARY:
Lipoprotein (a) [Lp (a)] is an independent cardiovascular risk (CVR) both in the general population and in patients with type 2 diabetes mellitus (DM-2). Until now no effective treatment is known to decrease the levels of Lp (a) levels and thus achieve a reduction of CVR. Among the new antidiabetic drugs are GLP-1Receptor agonists(GLP-1R). In addition to lowering blood glucose, these drugs have other beneficial effects. In our laboratory we have demonstrated that both native GLP-1 and various GLP-1R agonsits reduce the synthesis of Lp (a) in hepatocytes. The objective of the study is to test in humans the results observed in vitro. We will analyze whether treatment with GLP-1R agonists (Liraglutide, Exenatide or Lixisenatida) will reduce serum levels of Lp (a) in patients with DM-2.

DETAILED DESCRIPTION:
Background: Lipoprotein (a) [Lp (a)] is an independent cardiovascular risk (CVR) both in the general population and in patients with type 2 diabetes mellitus (DM-2). Until now no effective treatment is known to decrease the levels of Lp (a) levels and thus achieve a reduction of CVR. Among the new antidiabetic drugs are GLP-1Receptor agonists(GLP-1R). In addition to lowering blood glucose, these drugs have other beneficial effects. In our laboratory we have demonstrated that both native GLP-1 and various GLP-1R agonsits reduce the synthesis of Lp (a) in hepatocytes.

Hypothesis: Treatment with GLP-1R agonists will lower the levels of Lp (a) in patients with DM-2.

Objective: The objective of the study is to confirm in humans the results observed in vitro. We will analyze whether treatment with GLP-1R agonists (Liraglutide, Exenatide or Lixisenatida) will reduce serum levels of Lp (a) in patients with DM-2.

Methods: we will evaluate 40 patients with DM-2 treated at the Endocrinology Department of the Vall d'Hebron University Hospital. The patients will be distributed in two groups according to the treatment prescribed by the endocrinologist during the visit of routine monitoring: group A (20 patients who were prescribred treatment with GLP-1R agonists) and group B (20 patients who were not prescribed this treatment). According to the current guidelines for treating DM-2, the GLP-1R agonists are situated as a second line treatment after metformin, and the treatment should be individualized according to the characteristics of each patient. (Inzucchi et al. Management of hyperglycemia in type 2 diabetes: a patient-centered approach: position statement of the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD) Diabetes Care 2012; 35 (6):.. 1364-1379). Following these recommendations, the GLP-1R agonists are usually selected when there is obesity and / or very important to avoid hypoglycaemia. The decision to prescribe a GLP-1R agonist is made by the endocrinologist before and independently of the patient´s participation in the study.

Blood levels of Lp(a) will be evaluated at baseline and at 2 months (+/- 15 days). Diabetic patients who are treated with insulin, enzyme inhibitors DPP-4 (IDDP-4) or already treated with receptor agonists GLP-1, presenting with kidney and liver failure, HbA1c> 10%, LDL-cholesterol> 180 mg / dl and / or triglycerides> 350 mg / dl will excluded.

Relevance: The results will identify a potential treatment for lowering levels of Lp (a) in patients with DM-2 and thus reducing cardiovascular risk associated with this lipoprotein.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* age between 50-65 years
* written informed consent

Exclusion Criteria:

* active GLP-1R agonist, insulin or DPP-IV treatment.
* Liver failure (3lsn AST and/or ALT)
* Kidney failure (FG <30ml/min/1,73m2),
* HbA1c> 10%
* LDL-cholesterol> 180 mg/dl
* Triglycerides> 350 mg/dl

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-07 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Change in blood levels of Lipoprotein (a) (Lp(a)) | Baseline and two months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Hernandez C, Francisco G, Chacon P, Simo R. Lipoprotein(a) as a risk factor for cardiovascular mortality in type 2 diabetic patients: a 10-year follow-up study. Diabetes Care. 2005 Apr;28(4):931-3. doi: 10.2337/diacare.28.4.931. No abstract available. PMID 15793200
- [Background] Hernandez C, Francisco G, Chacon P, Mesa J, Simo R. Biological variation of lipoprotein(a) in a diabetic population. Analysis of the causes and clinical implications. Clin Chem Lab Med. 2003 Aug;41(8):1075-80. doi: 10.1515/CCLM.2003.166. PMID 12964817
- [Background] Genser B, Dias KC, Siekmeier R, Stojakovic T, Grammer T, Maerz W. Lipoprotein (a) and risk of cardiovascular disease--a systematic review and meta analysis of prospective studies. Clin Lab. 2011;57(3-4):143-56. PMID 21500721